CLINICAL TRIAL: NCT05180045
Title: Home Blood Pressure Telemonitoring LINKED With Community Health Workers to Improve Blood Pressure
Acronym: LINKED-BP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00307545
Record Dates: First submitted 2021-12-14; First posted 2022-01-06 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LINKED-BP Program (Experimental): Patients in the LINKED-BP Program will be trained to measure their BP with an Omron 10 series device. Patients who have smartphones will download the patient facing app and receive a unique link from the study team. Patients who do not own a smartphone will be provided one with a data plan for the duration of the study. The primary care provider and CHW will be able to visualize the remotely transmitted data via the clinician portal.
  CHWs will support patients by: (1) providing education on how to manage BP through self-monitoring and practicing dietary modification and exercise; (2) reinforcing positive BP self-management through follow-up encounters; (3) assisting with linkages to existing clinical and administrative services; and (4) link participants with community resources to address health-related social needs.
  The staff in each participating community health center practice will be trained in blood pressure measurement best practices.
  Interventions: Behavioral: LINKED-BP Program
- Enhanced Usual Care (No Intervention): Patients in the Enhanced Usual Care Arm, will receive care as usual from thier primary care provider and will be trained to measure their BP with an Omron 10 series device. The staff in each participating community health center practice will be trained in blood pressure measurement best practices.

INTERVENTIONS:
Behavioral: LINKED-BP Program — The intervention arm will include training on HBPM, Sphygmo BP telemonitoring app, and CHW visits for education and counseling on lifestyle modification. Patients will be trained to measure their BP in the morning and evening for 7 days. Patients enter data using Bluetooth device transmission or manual entry. Guidance is provided on accurate BP measurement. The app stores and securely relays data to the cloud. The primary care provider and CHW will be able to visualize the remotely transmitted data via the clinician portal. Other components of usual care at the practices may include dietary counseling, on-site clinical pharmacists, social workers, case managers as needed for BP follow up, and assistance with medications and appointments as needed. The intervention period for each study participant is 12 months.
  Arms: LINKED-BP Program

SUMMARY:
The LINKED-BP Program is a patient-centered, multi-level intervention linking home blood pressure monitoring (HBPM) with a telemonitoring platform (Sphygmo) that links with all Bluetooth-enabled validated blood pressure (BP) devices, support from community health workers (CHWs), and BP measurement training at community health centers serving high-risk adults to prevent stage 2 hypertension (BP ≥ 140/90 mm Hg). The LINKED-BP Program study will recruit a total of 600 adults (30 from each practice) with elevated BP (120-129/<80 mm Hg) or untreated stage 1 hypertension (130-139/80-89 mm Hg) across 20 community health centers or primary care practices serving high-risk adults. This cluster-randomized trial consists of two arms: (1) enhanced "usual care arm," wherein patients will be provided with Omron 10 series home BP monitors (HBPM) and will be managed by the patients' primary care clinicians as usual; and (2) the LINKED-BP Program or "intervention arm," which will include training of patients on HBPM, Sphygmo BP telemonitoring app, and CHW visits for education and counseling on lifestyle modification. The intervention period for each study participant is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age as of the date of data extraction
* Self-identify as non-Hispanic white, non-Hispanic African-American or Hispanic
* Have elevated BP (120-129/<80 mm Hg) or untreated stage 1 hypertension (130-139/80-89 mm Hg) (defined by AHA's 2017 hypertension clinical guidelines)
* Receives primary medical care at one of the participating community health centers and primary care practices

Exclusion Criteria:

* Age <18 years
* Prescribed antihypertensive medication
* Diagnosis of end-stage renal disease (ESRD)
* Condition which interferes with outcome measurement (e.g., dialysis)
* Serious medical condition which either limits life expectancy or requires active management (e.g., cancer)
* Patients with serious cognitive impairment or other conditions preventing their participation in the intervention
* Upper arm circumference >50 cm (maximum limit of the extra-large BP cuff)
* Those planning to leave the practice or move out of the geographic area in 18 months
* Those who no longer consider the practice site the location where they receive primary care
* Unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Baseline and 12 months
  Change in systolic blood pressure in millimeters of mercury (mmHg) over a 12 month period.

SECONDARY OUTCOMES:
Change in diastolic blood pressure | Baseline and 12 months
  Change in diastolic blood pressure in millimeters of mercury (mmHg) over a 12 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Commodore-Mensah, PhD, MHS, RN, Principal Investigator — JHU School Of Nursing
Locations (20):
- United States (20):
  - Johns Hopkins Community Physicians I Street, Washington D.C., District of Columbia
  - Unity Upper Cardozo Health Center, Washington D.C., District of Columbia
  - Unity Brentwood Health Center, Washington D.C., District of Columbia
  - Unity East of the River, Washington D.C., District of Columbia
  - Unity Minnesota Avenue Health Center, Washington D.C., District of Columbia
  - Unity Parkside Health Center, Washington D.C., District of Columbia
  - Unity Anacostia Health Center, Washington D.C., District of Columbia
  - Johns Hopkins Community Physicians Remington, Baltimore, Maryland
  - Johns Hopkins Community Physicians Bowie, Bowie, Maryland
  - Johns Hopkins Community Physicians Brandywine, Brandywine, Maryland
  - Choptank Fassett Magee Medical and Cambridge Dental Center, Cambridge, Maryland
  - Choptank Denton Health Center, Denton, Maryland
  - Johns Hopkins Community Physicians Greater Dundalk, Dundalk, Maryland
  - Choptank Easton Health Center, Easton, Maryland
  - Choptank Federalsburg Medical and Dental Center, Federalsburg, Maryland
  - Johns Hopkins Community Physicians Fulton, Fulton, Maryland
  - Choptank Goldsboro, Goldsboro, Maryland
  - Johns Hopkins Community Physicians White Marsh, Nottingham, Maryland
  - Choptank Bay Hundred, Saint Michaels, Maryland
  - Johns Hopkins Community Physicans Charles County-White Plains, White Plains, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Commodore-Mensah Y, Liu X, Ogungbe O, Ibe C, Amihere J, Mensa M, Martin SS, Crews D, Carson KA, Cooper LA, Himmelfarb CR. Design and Rationale of the Home Blood Pressure Telemonitoring Linked with Community Health Workers to Improve Blood Pressure (LINKED-BP) Program. Am J Hypertens. 2023 Apr 15;36(5):273-282. doi: 10.1093/ajh/hpad001. PMID 37061796